CLINICAL TRIAL: NCT02866422
Title: Development of an Instrument That Monitors Behaviors Associated With OCD
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Collaborators: U.S. National Science Foundation (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 1403M49006; CNS 1338042 (Other Grant/Funding Number: United States National Science Foundation)
Record Dates: First submitted 2016-08-01; First posted 2016-08-15 (Estimated); Last update posted 2016-08-15 (Estimated); Status verified 2016-08

CONDITIONS: OCD
Keywords: OCD

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- OCD
  Interventions: Other: No Intervention
- Healthy Controls
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — Observational Study: No intervention

SUMMARY:
To support the discovery of new means for revealing the presence of Obsessive Compulsive Disorder (OCD), facilitating detection through new technology-based metrics, and attempt to automate existing diagnostic procedures allowing for more efficient diagnostic methods that would broaden clinical scope and outreach.

DETAILED DESCRIPTION:
Aim 1: To observe and compare childhood behaviors regarding handwashing in OCD and control populations

Hypothesis 1: Control participants will spend less time washing their hands, will wash them less frequently, and will be less preoccupied with the sink when doing other activities.

Aim 2: To observe and compare childhood behaviors regarding organizing a cluttered area.

Hypothesis 2: OCD participants will be more disturbed by the presence of clutter and more compelled to organize the items than control participants

Aim 3: To observe and compare childhood behaviors regarding turning on/off light switches

Hypothesis 3: OCD children will be more likely to exhibit compulsive repetitive behaviors regarding the light switch than control participants

ELIGIBILITY:
Inclusion Criteria:

* Male and female children
* Aged 5 to 17

Exclusion Criteria:

* Inability or unwillingness to provide written informed consent/assent

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The investigators will recruit 20 children and adolescents with OCD aged 5-17 who present to the University of Minnesota Child and Adolescent Anxiety and Mood Disorders Clinic or who are referred from outside clinicians. Twenty healthy controls will be recruited from the community.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2014-03; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Length of Handwashing | Same Day
  Researchers blindly rate the how long (secs) it takes participants to wash their hands.
Behaviors Associated with Handwashing | Same Day
  Researchers blindly rate whether participants exhibit any unique behavior while washing their hands.
Length of Free Arrangement | Same Day
  Researchers blindly rate how long it takes participants to freely organize a box of school supplies.
Frequency of Movements During Free Arrangement | Same Day
  Researchers blindly rate how many times participants move an object while freely arranging a box of school supplies.
Amount of Space Used During Free Arrangement | Same Day
  Researchers blindly rate how much space participants use while freely arranging a box of school supplies (small, medium, or large space).
Length of Carpet Arrangement | Same Day
  Researchers blindly rate and compare how long (secs) it takes participants to arrange a box of school supplies on a plain versus patterned carpet.
Frequency of Movements During Carpet Arrangement | Same Day
  Researchers blindly rate and compare how many times participants move an object while arranging a box of school supplies on a plain versus patterned carpet.
Frequency of Adjustments During Carpet Arrangement | Same Day
  Researchers blindly rate and compare how many times participants adjust the positioning of an object while arranging a box of school supplies on a plain versus patterned carpet.
Size of Arrangement According to Sample | Same Day
  Researchers blindly rate and compare how accurately participants replicate the size of the arrangement according to a sample picture (smaller than sample, approximate to sample, larger than sample) on a plain versus patterned carpet.
Frequency of Checking the Sample | Same Day
  Researchers blindly rate and compare how many times participants check the sample picture of the arrangement while organizing a box of school supplies on a plain versus patterned carpet.

CONTACTS AND LOCATIONS:
Overall Officials: Gail A Bernstein, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Bernstein GA, Hadjiyanni T, Cullen KR, Robinson JW, Harris EC, Young AD, Fasching J, Walczak N, Lee S, Morellas V, Papanikolopoulos N. Use of Computer Vision Tools to Identify Behavioral Markers of Pediatric Obsessive-Compulsive Disorder: A Pilot Study. J Child Adolesc Psychopharmacol. 2017 Mar;27(2):140-147. doi: 10.1089/cap.2016.0067. Epub 2016 Nov 10. PMID 27830935